CLINICAL TRIAL: NCT02067104
Title: A Placebo Controlled Double-Blind Study to Evaluate the Efficacy of Vismodegib as Chemoprevention of New Bcc Development in High Risk Subjects
Brief Title: Vismodegib in Basal Cell Carcinomas (BCC) Chemoprevention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1401183410; ML28585 (Other: Genentech BioOncology)
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Basal Cell Carcinomas
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): receive 150 mg of oral placebo daily for a period of 2 months
  Interventions: Drug: Placebo
- Vismodegib (Experimental): receive 150 mg of vismodegib daily for a period of 2 months
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — Pulse therapy pattern of 2 months of daily treatment and 2 months of no treatment for 24 months.
  Other Names: Erivedge
  Arms: Vismodegib
Drug: Placebo — Pulse therapy pattern of 2 months of daily treatment and 2 months of no treatment for 24 months.
  Arms: Placebo

SUMMARY:
This study is a single site double blinded Phase II study to evaluate the chemopreventative effectiveness of vismodegib in the treatment of subjects at high risk for developing basal cell carcinomas (BCC).

DETAILED DESCRIPTION:
The primary objective of this study will be to determine if vismodegib pulse therapy will significantly reduce the incidence of newly diagnosed basal cell carcinomas (BCC) in high risk individuals when compared with placebo, as measured by the incidence of biopsy confirmed BCC over a 24 month period.

The secondary objective will be to determine that there will be no difference in the incidence of newly diagnosed squamous cell carcinomas (SCC) in the same subjects receiving vismodegib treatment when compared with placebo, as measured by the incidence of biopsy confirmed SCC over the same 24 month period.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects
* Comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* At least 18 years of age at the time of informed consent.
* History of 3 or more biopsy confirmed BCCs in the preceding 2 years, calculated from 2 years prior to the screening visit.
* No active skin cancers.
* Women of reproductive potential must agree to use two forms of acceptable contraception
* Male subjects must agree to use condoms at all times, even after a vasectomy, during sexual intercourse with female partners of reproductive potential during treatment with vismodegib and for 2 months after the last dose to avoid exposing a pregnant partner and the unborn fetus to vismodegib.
* Male patients must agree not to donate sperm during the study and for 2 months after discontinuation of vismodegib
* Agreement not to donate blood or blood products during the study and for 7 months after the last dose.
* Ability to understand and the willingness to sign a written informed consent document in English

Exclusion Criteria:

* Women who are pregnant or lactating, or planning pregnancy while enrolled in the study or for 7 months after the last dose of the study drug.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Subjects with clinically stable chronic medical conditions including, but not limited to, controlled hypertension, diabetes mellitus type II, hypercholesterolemia, or osteoarthritis, will be allowed to enter the study.
* Inability or unwillingness to swallow capsules.
* Have a history of alcohol of substance abuse, unless in full remission for greater than 6 months prior to the screening visit (Day 0) when the consent form is signed.
* Known to be infected with human immunodeficiency virus (HIV), hepatitis B or hepatitis C viruses.
* Currently receiving vismodegib, biologics or chemotherapy
* Currently undergoing treatment with photodynamic therapy, topical chemotherapy agents including Imiquimod, fluorouracil
* Subjects who have Gorlins syndrome
* Subjects who have received any type of solid organ transplant
* Subjects taking immunosuppressive medications at the screening visit. (Day 0)
* Participation in other study using an investigational or experimental therapy or procedure within 4 weeks or 5 half-lives (whichever is longer) before the screening visit and/or during study participation. Subjects cannot participate in studies of other investigational or experimental therapies or procedures at any time during their participation in this study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects unable or unwilling to comply with the study visit schedule and requirements of the study
* Subjects unable to speak and read the English language
* A subject who, in the opinion of the sponsor-investigator will be uncooperative or unable to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Curiel-Lewandroski, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vismodegib
Started | 4 | 5
Completed | 0 | 0
Not Completed | 4 | 5
Not completed — Study termination due to low accrual | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vismodegib | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Vismodegib Pulse Therapy on the Incidence of Newly Diagnosed Basal Cell Carcinomas (BCC)
Description: Measured by the incidence of biopsy confirmed BCC over a 24 month period
Time Frame: 24 Months
Population: Early study termination due to low accrual. No data analyzed; no results.
Arm/Group | Placebo | Vismodegib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Incidence of Newly Diagnosed Squamous Cell Carcinomas (SCC) in the Same Subjects Receiving Vismodegib Treatment When Compared With Placebo
Description: Measured by the incidence of biopsy confirmed SCC over the same 24 month period
Time Frame: 24 Months
Population: Early study termination due to low accrual. No data analyzed; no results.
Arm/Group | Placebo | Vismodegib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Vismodegib
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | Vismodegib (N=5)
Scale in ear (Skin and subcutaneous tissue disorders) | 0 | 1
Taste disturbance (Gastrointestinal disorders) | 1 | 3
Leg cramps (Musculoskeletal and connective tissue disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes